CLINICAL TRIAL: NCT00749411
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, 4-week Study to Evaluate the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Repeat Inhaled Doses of the Combination of GSK233705 and GW642444 Administered Once-daily in Subjects With COPD
Brief Title: Safety and Tolerability of Repeat Dosing of GSK233705/GW642444 in COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DB1111581; NCT00843206 (obsolete NCT alias)
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; long-acting beta agonist; Emphysema; Chronic Bronchitis; Chronic Obstructive Pulmonary Disease (COPD); bronchodilator; long acting muscarinic antagonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: GSK233705/GW642444
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — matching placebo
  Arms: Arm 2
Drug: GSK233705/GW642444 — The combination of the long-acting muscarinic antagonist GSK233705 and the long acting beta agonist GW642444 in a single inhaler.
  Arms: Arm 1

SUMMARY:
The purpose of this study is the evaluate the safety and tolerability of repeat dosing of the combination of inhaled GSK233705 and GW642444 administered once-daily in subjects with COPD.

ELIGIBILITY:
Inclusion Criteria:

* male and females 40 to 80 years of age (inclusive)
* COPD diagnosis
* Current or previous smokers with a cigarette smoking history of at least 10 pack-
* Post-albuterol FEV1/FVC of 0.70 or less
* Post-albuterol FEV1 of 35% to 80% (inclusive)

Exclusion Criteria:

* Pregnant or lactating females
* current diagnosis of asthma
* respiratory disorders other than COPD
* clinically significant cardiovascular, neurological, psychiatric, renal, immunological, endocrine, or hematological abnormalities that are uncontrolled
* clinically significant sleep apnea
* previous lung resection surgery
* clinically significant abnormalities confirmed by chest x-ray that are not related to COPD
* hospitalization for COPD within 3 months of screening
* use of antibiotics for lower respiratory tract infection within 6 months of screening
* abnormal and clinically significant 12-lead ECG findings
* current malignancy in remission for less that 5 years
* medical conditions that would contraindicate the use of anticholinergics
* positive hepatitis B or C test
* history of alcohol or drug abuse
* unable to withhold albuterol for 6 or more hours
* use of long term oxygen therapy
* conditions that would limit the validity of informed consent
* use of GW642444 or GSK233705 in previous studies
* use of an investigation drug with 30 days of screening
* use of inhaled corticosteroids (ICS) at a dose greater than 1000mcg of fluticasone propionate or equivalent
* hypersensitivity to beta-agonists
* concurrent use of long-acting beta-agonists (LABA) or long-acting muscaring antagonists, LABA/ICS combination products, cytochrome p450 inhibitors, oral or depot corticosteroids, theophyllines, oral beta agonists, oral leukotrine modulators, inhaled short acting anticholinergics.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-11-13 (Actual); Primary Completion 2009-02-12 (Actual); Study Completion 2009-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- United States (12):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Biddeford, Maine
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Summit, New Jersey
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] GSK has submitted manuscripts of these study results to peer-reviewed scientific journals which were not accepted for publication. GSK is providing the attached study results summary with a conclusion.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: DB1111581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: DB1111581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: DB1111581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: DB1111581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: DB1111581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: DB1111581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: DB1111581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between 13 November 2008 and 12 February 2009, at 12 centers in the United States.
Pre-assignment Details: A total of 127 participants were screened out of which 61 participants were enrolled and randomized to receive at least one dose of study medication in the study.
Groups:
- Placebo: Eligible participants received oral inhalation of matching Placebo via dry powder inhaler (DPI) once daily for 28 days.
- GSK233705/GW642444: Eligible participants received oral inhalation of GSK233705 100 microgram (mcg)/GW642444 25 mcg via DPI once daily for 28 days.
Period: Overall Study
Arm/Group | Placebo | GSK233705/GW642444
Started | 21 | 40
Completed | 20 | 35
Not Completed | 1 | 5
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Protocol-defined stopping criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Eligible participants received oral inhalation of matching Placebo via DPI once daily for 28 days.
- GSK233705/GW642444: Eligible participants received oral inhalation of GSK233705 100 mcg / GW642444 25 mcg via DPI once daily for 28 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK233705/GW642444 | Total
Number analyzed (Participants) | 21 | 40 | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (10.09) | 61.2 (9.55) | 61.0 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 11 | 29 | 40
Race/Ethnicity, Customized [Number; unit: Participants]
  African American / African Heritage | 0 | 2 | 2
  Asian - East Asian Heritage | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 20 | 38 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weighted Mean Pulse Rate Over (0-4 Hours) at Day 28.
Description: Baseline was the most recent result taken on or before pre-dose (Day 1). The analysis was performed using a Repeated Measures Model. This model used all available weighted mean pulse rate values recorded. Change from Baseline was calculated as (Change from Baseline = Assessment value - Baseline value).
Time Frame: Baseline (Pre-dose, Day 1) and Day 28
Population: Intent-to-Treat (ITT) Population comprised of all participants who were randomized to study treatment and took at least one dose of study medication. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Beat per minute (bpm)
Arm/Group | Placebo | GSK233705/GW642444
Number analyzed (Participants) | 20 | 35
Beat per minute (bpm) | -3.8 (1.78) | -4.8 (1.32)
Statistical Analysis 1: Comparison: Placebo vs GSK233705/GW642444; Test type: Non-Inferiority — GSK233705/GW642444 were declared non-inferior to placebo for heart rate if the upper limit of the 95% confidence interval for the estimated treatment difference for weighted mean heart rate was less than +10bpm; Mean Difference (Net) = -1.0, 95% CI 2-sided [-5.5 to 3.5] — Analysis performed using a Repeated Measures Model with covariates of baseline pulse rate, sex, age, smoking status, treatment and Day and Day by treatment and Day by baseline interactions

2. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE was defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE include AEs those result in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: On-treatment; from treatment start until one day after treatment stop (Up to Day 29)
Population: ITT Population.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK233705/GW642444
Number analyzed (Participants) | 21 | 40
Participants
  Any AE | 8 | 10
  Any SAE | 0 | 0

ADVERSE EVENTS:
Time Frame: On-treatment; from treatment start until one day after treatment stop (Up to Day 29)
Description: Intent to treat population was used to collect the AEs. There were no on-treatment SAEs reported in the study. Only on-treatment SAEs and nSAEs are presented.
Arm/Group | Placebo | GSK233705/GW642444
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/40
Other Adverse Events (participants affected / at risk) | 8/21 | 10/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=21) | GSK233705/GW642444 (N=40)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.